CLINICAL TRIAL: NCT04106284
Title: Comorbidities of Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, hasnaa abdalla, resident doctor, Assiut University
Other Study IDs: Comorbidities of epilepsy
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epilepsy is the second commonest chronic neurological disorder in developed countries, Comorbidity refers to the co-occurrence of two conditions with a greater frequency than found in the general population

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed as primary epilepsy either newly diagnosed or on AEDs
* Aged above 18 years old
* Males and females

Exclusion Criteria:

* Patients diagnosed as secondary epilepsy (post stroke, trauma, tumor, encephalitis, etc).
* Patients diagnosed as epilepsy syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included will be chosen from Epilepsy out patient clinic and Neurology department at Assiut University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-01 (Estimated)

PRIMARY OUTCOMES:
DEXA Scan | 1 year
  DEXA scan to measure bone mineral density at 3 points (wrist joint ,hip joint and lumbo-sacral vertebrae)